CLINICAL TRIAL: NCT00434590
Title: Controlled, Randomized, Parallel Group Study to Assess Efficacy and Tolerability of Full Dose Enteric-coated Mycophenolate Sodium, in Addition to Cyclosporine for Microemulsion Reduced Dose, in Maintenance Renal Transplant Recipients
Brief Title: Efficacy and Tolerability of Full Dose Enteric-coated Mycophenolate Sodium, in Addition to Cyclosporine for Microemulsion Reduced Dose, in Maintenance Renal Transplant Recipients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study has been stopped because of the lack of enrollment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CERL080AIT09
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Results first posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-03

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Mycophenolic Acid; Immunosuppression; Cyclosporine
MeSH Terms: interventions — Mycophenolic Acid

ARMS (2):
- Full Dose Myfortic® and Reduced Dose Neoral® (Experimental): The administration of gradual dose increased to reach 1440 mg/day (V4) of enteric-coated mycophenolate sodium (Myfortic®, EC-MPS) with simultaneous dose reduction of micro emulsion cyclosporine (Neoral®, CsA-ME) given to maintenance kidney transplant patients previously treated with reduced-dose mycophenolate mofetil (MMF) and standard dose CsA-ME
  Interventions: Drug: Enteric coated mycophenolate sodium (Myfortic®)
- Standard Dose of Myfortic® and Standard Dose of CsA-ME (Active Comparator): Patients received unchanged dose of Myfortic® (equimolar to the prior established dose MMF) and unchanged standard dose of CsA-ME.
  Interventions: Drug: Enteric coated mycophenolate sodium (Myfortic®)

INTERVENTIONS:
Drug: Enteric coated mycophenolate sodium (Myfortic®)
  Other Names: Myfortic

SUMMARY:
The study will evaluate kidney graft function in maintenance renal transplant patients.

ELIGIBILITY:
Inclusion criteria:

* Male or female recipients of single or double renal transplant performed since at least one year and no more that 5 years
* Age > 18 yrs
* Adequate and stable renal function
* Informed consent.

Exclusion criteria:

* Kidney transplant combined with other organs;
* Significant proteinuria
* Severe ongoing infections;
* Present or historical malignant neoplasia, of any type, with the exception of excised non metastatic non-melanoma skin cancer and previous malignant neoplasia cured since at least 5 years;
* Relapse of the end-stage renal disease on the transplanted kidney;
* Leucopenia, thrombocytopenia or severe anemia;

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigative Site, Bologna, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Full Dose Myfortic® and Reduced Dose Neoral® | Standard Dose of Myfortic® and Standard Dose of CsA-ME
Started | 5 | 5
Completed | 0 (All patients randomized had study discontinued because of premature study termination.) | 0
Not Completed | 5 | 5
Not completed — Administrative problems | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Dose Myfortic® and Reduced Dose Neoral® | Standard Dose of Myfortic® and Standard Dose of CsA-ME | Total
Number analyzed (Participants) | 5 | 5 | 10
Age Continuous [Mean (Standard Deviation); unit: Years] | 52.4 (13.8) | 58.0 (12.5) | 55.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Renal Function, as Assessed by Glomerular Filtration Rate (GFR) at 12 Months
Description: The 12 month change from baseline (visit 2) in the glomerular filtration rate using the abbreviated Modification of Diet in Renal Disease (MDRD) formula to calculate GFR using the participant's serum creatinine, age, gender and ethnicity.
Time Frame: 12 months
Population: Study was terminated without analysis (small sample size).
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Full Dose Myfortic® and Reduced Dose Neoral® | Standard Dose of Myfortic® and Standard Dose of CsA-ME
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Creatinine Clearance at 12 Months
Time Frame: 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Serum Creatinine at 12 Months
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Reciprocal Slope of Serum Creatinine (mg/dL) or Micromole/l at 12 Months
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Biopsy Proven Acute Rejections and Clinically Confirmed Acute Rejection at 12 Months
Time Frame: 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Chronic Rejection as Confirmed by Renal Biopsy at 12 Months
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Full Dose Myfortic® and Reduced Dose Neoral® | Standard Dose of Myfortic® and Standard Dose of CsA-ME
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Full Dose Myfortic® and Reduced Dose Neoral® (N=5) | Standard Dose of Myfortic® and Standard Dose of CsA-ME (N=5)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Conjunctival irritation (Eye disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.